CLINICAL TRIAL: NCT05019495
Title: Optimizing Tobacco Treatment Delivery for People Living With HIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alana Rojewski, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00107332; R01CA261232 (NIH)
Record Dates: First submitted 2021-05-04; First posted 2021-08-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Hiv; Smoking, Cigarette
Keywords: Smoking
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cigarette Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Treatment as Usual (TAU) participants will follow traditional clinic pathways for receiving tobacco treatment in the Medical University of South Carolina Health Infectious Disease outpatient clinic. All patients randomized to TAU will have the opportunity to access smoking cessation pharmacotherapy from the Infectious Disease clinical pharmacist.
- ProMOTE (Experimental): In the PrOMOTE group, the participants will be contacted by the clinical pharmacist on the tobacco treatment staff three times for medication prescriptions and refills. They will also receive brief counseling and motivational interviewing by the clinical pharmacist.
  Interventions: Behavioral: PrOMOTE

INTERVENTIONS:
Behavioral: PrOMOTE — This is an opt-out, proactive approach to tobacco treatment by a clinical pharmacy specialist. The pharmacist will call patients and offer an individualized pharmacotherapy prescription. The patient must opt-out for it not to be sent to their pharmacy. The patient will also receive brief motivational interviewing and behavioral counseling from the pharmacist.
  Other Names: Proactive Outreach with Medication Opt-out for Tobacco Treatment Engagement
  Arms: ProMOTE

SUMMARY:
The purpose of this study is to conduct a randomized trial to evaluate a proactive, opt-out model of provider contact to deliver smoking cessation support for people living with HIV compared to standard care support delivered through traditional clinic pathways. Investigators will also evaluate implementation outcomes to identify barriers and facilitators towards future implementation. Investigators hope to define best practices and optimize the delivery of smoking cessation interventions for people living with HIV.

DETAILED DESCRIPTION:
This hybrid effectiveness-implementation trial presents on opportunity to optimize tobacco treatment delivery for people living with HIV (PLWH), and identify barriers and facilitators towards future implementation. We are proposing a comparison of Treatment As Usual (TAU; reactive, opt-in tobacco treatment using standard clinical pathways) vs Proactive Outreach with Medication Opt-out for Tobacco Treatment Engagement (PrOMOTE). Participants will be randomized in a 1:1 allocation. The primary aim is to compare rates of cessation and quit attempts at the Week 12 follow-up between participants who received TAU versus PrOMOTE. As a secondary aim we will characterize key determinants of PrOMOTE reach, implementation fidelity, adherence, and acceptability. We hypothesize that the PrOMOTE intervention will increase cessation rates and number of quit attempts, and that it will result in greater reach and pharmacotherapy delivery compared to TAU. Key determinants of PrOMOTE implementation outcomes will also be characterized. An exploratory assessment of CD4 cell count and HIV viral load, in addition to durability of smoking cessation outcomes, will also be assessed. By optimizing the delivery of effective tobacco treatments for PLWH, we hope to increase the number of people receiving tobacco treatment, increase tobacco cessation rates, and reduce the risk of morbidity and mortality from smoking-related causes.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 and older
* Current diagnosis of HIV
* Current smoker (defined as self-report of current smoking)
* Willing to be randomized
* English speaking

Exclusion Criteria:

* Currently taking part in any other tobacco treatment program or using cessation medication (i.e., taking nicotine replacement therapy or other cessation medications, enrolled in the Quitline, or in another study)
* Currently imprisoned
* Pregnant women
* Non-English speaking persons

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Tobacco use abstinence | 7 days
  Self-reported and confirmed by breath carbon monoxide test

SECONDARY OUTCOMES:
Reach | 24 weeks (study completion)
  Percentage of current smokers engaged in an intervention
Fidelity of intervention | 24 weeks (study completion)
  The extent to which an intervention is implemented as intended. This will be collected via interviews with patients and providers.
Fidelity of intervention | 24 weeks (study completion)
  The extent to which an intervention is implemented as intended. This will be collected via surveys.
Perceived barriers to the outcomes | 24 weeks (study completion)
  Using the implementation tracking checklist, provider perceptions of barriers faced in completion of intervention steps will be monitored. These will be collected via interviews with patients.
Perceived barriers to the outcomes | 24 weeks (study completion)
  Using the implementation tracking checklist, provider perceptions of barriers faced in completion of intervention steps will be monitored. These will be collected via interviews with providers.
Acceptability of intervention | 24 weeks (study completion)
  The perception among stakeholders that the treatment is agreeable or satisfactory. This will be collected via interviews with patients and providers.
Acceptability of intervention | 24 weeks (study completion)
  The perception among stakeholders that the treatment is agreeable or satisfactory. This will be collected via surveys.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanford BT, Toll BA, Eckard AR, Sterba KR, Cummings KM, Baker NL, Rojewski AM. Optimizing tobacco treatment delivery for people with HIV: trial protocol for a randomized controlled trial. Addict Sci Clin Pract. 2022 Nov 5;17(1):61. doi: 10.1186/s13722-022-00341-2. PMID 36335376